CLINICAL TRIAL: NCT05794711
Title: Concordance Between Intraoperative Frozen Section Pathology and Postoperative Paraffin-embedded Pathology in Diagnosing the IASLC Grade of Lung Adenocarcinoma
Brief Title: Intraoperative Frozen Section Pathology to Guide Surgical Treatment for Lung Adenocarcinoma (ECTOP-1015)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Other Study IDs: CONCORD-B
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Lung Adenocarcinoma; Surgical Procedure, Unspecified; Pathology
Keywords: Intraoperative frozen section pathology; Surgical treatment; Lung adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical T1N0M0 lung adenocarcinoma patients eligible for surgery.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection of lung adenocarcinoma. Wedge resection, segmentectomy or lobectomy will be performed according to each patients' condition.

SUMMARY:
This study is one of Eastern Cooperative Thoracic Oncology Projects (ECTOP-1015). The goal of this clinical trial is to confirm the concordance rate between intra-operative frozen section pathological diagnosis and post-operative paraffin embedded pathological diagnosis, and use this result to guide surgical treatment for early stage (cT1N0M0) lung adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent form and are willing to complete the study according to the study protocol;
* No previous history of cancer or pulmonary surgery;
* Solitary lesions or multiple lesions with only one not manifesting as pure ground-glass opacity (GGO) on CT scan;
* Peripheral clinical T1N0M0 patients that are eligible for surgery;
* Non-small cell lung cancer is pathologically diagnosed before or at surgery;
* No radiation therapy or chemotherapy before surgery.

Exclusion Criteria:

* Patients with clinical stages other than T1N0M0;
* The lesion cannot be completely resected;
* Previous history of cancer;
* Patients having received radiation therapy or chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical stage T1N0M0 lung adenocarcinoma patients who are going to undergo surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of IASLC grades of lung adenocarcinoma

SECONDARY OUTCOMES:
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of lung adenocarcinoma subtypes according to the WHO classifications.
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of pleural invasion and lymph node invasion.
Concordance rate | 2 years
  Concordance rate between intraoperative frozen section and postoperative paraffin embedded pathology in making the diagnosis of spread through air space (STAS).
Recurrence-free survival (RFS) | 5 years
  Recurrence-free survival (RFS) is defined as the time from date of curative surgery to the time of recurrence or death, whichever comes first.
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the time from date of curative surgery to the time of death of any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fu Z, Shen X, Deng C, Cao H, Jin Y, Zheng Q, Yang Y, Qian B, Yuan C, Wang W, Zhang L, Song Q, Zuo S, Ma J, You S, Zheng S, Gao Q, Su G, Zhang Y, Fu F, Chen H, Li Y. Prediction of the pathological subtypes by intraoperative frozen section for patients with cT1N0M0 invasive lung adenocarcinoma (ECTOP-1015): a prospective multicenter study. Int J Surg. 2024 Sep 1;110(9):5444-5451. doi: 10.1097/JS9.0000000000001667. PMID 38781043